CLINICAL TRIAL: NCT02308371
Title: Automated Pulse Pressure Variation Guided Fluid Management in the Pediatric Intensive Care Setting
Brief Title: PPV to Guide Fluid Management in the PICU
Acronym: PPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-2019
Record Dates: First submitted 2014-10-24; First posted 2014-12-04 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-06

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome
Keywords: critically ill pediatric patients; fluid resuscitation
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective (Experimental): Patients in this arm will have fluid given based on standard clinical data (blood pressure, heart rate, lactate level, urine output) in addition to information provided by automated pulse pressure variation (PPV). PPV will be followed for first 48 hours after recruitment to the study. Fluid (normal saline, albumin 5%, hetastarch per the clinician preference) will be given in 5cc/kg increments for PPV> 13 (in addition to standard clinical data) until PPV < 13.
  Interventions: Device: Automated Pulse Pressure Variation
- Retrospective (No Intervention): Patients in this arm were previously admitted to the PICU and were given fluid based on standard clinical data. PPV was not used to guide therapy in this group of patients.

INTERVENTIONS:
Device: Automated Pulse Pressure Variation — Based on standard of care, the physician will give fluid as needed based on standard clinical data (heart rate, central venous pressure if available, blood pressure, urine output, physical exam, lactate level) and pulse pressure variation. PPV should be elevated consistently greater than 15 minutes before giving fluid without other symptoms of patient instability (low blood pressure, elevated lactate, tachycardia). Pulse pressure variation will be followed for 48 hours.
  Other Names: Realtime automated pulse pressure variation algorithm; Philips MX800 monitor
  Arms: Prospective

SUMMARY:
Children who are critically ill often require large amounts of fluid during their acute illness. It has been shown in multiple studies that appropriate administration of fluid decreases morbidity and mortality, but giving too much fluid can also cause increased morbidity and mortality. It is often difficult to discern from physical exam, vital signs and labs if the amount of fluid that has been given is appropriate or if a pediatric patient requires more fluid. Pulse pressure variation (PPV) is the change in blood pressure when a patient is on a ventilator or breathing machine. PPV has been used in multiple adult studies to help predict fluid needs in a critically ill patient. In this study, we would like to investigate if PPV can help better predict if critically ill pediatric patients in the pediatric intensive care unit (PICU) need fluid. The investigators hope that by having the additional information that PPV can provide, physicians can more judiciously give fluid and thereby improve morbidity of critically ill patients in the PICU.

DETAILED DESCRIPTION:
In pediatric critical care, it is difficult to discern a patient's intravascular fluid status (hypovolemia, hypervolemia, euvolemia). Often, pediatric sepsis patients exhibit profound hypovolemia and early aggressive fluid resuscitation has been shown to decrease mortality (1,2). Within the first 48 hours of presentation, pediatric patients with sepsis can have profound changes in physiology with changes in cardiac function and systemic vascular resistance which can make it difficult to discern whether continued fluid resuscitation or the addition of vasopressor support is needed (1,2). Similar physiology can also be seen in other patients with systemic inflammatory response such as postoperative cardiac patients and general pediatric post-surgical patients. While appropriate fluid resuscitation is needed, it has been shown that fluid overload does increase mortality (3-5). Clinicians often use clinical exam, vital signs, urine output and central venous pressure (CVP) as guides for need of fluid resuscitation, but static measures such as central venous pressure, pulmonary wedge pressure, and clinical exam have not been shown to be strong predictors of fluid responsiveness and cardiac output in patients (6-8). A more accurate way to discern fluid status and heart function is through measurement of cardiac output, but in order to calculate cardiac output, additional tests such as an echocardiogram is needed or additional invasive monitoring using thermodilution such as a continuous cardiac output monitor is needed (7,8).

In the last 30 years, dynamic changes in arterial pressure during the respiratory cycle have been described, where there is a decrease in cardiac preload during time of inspiration of a positive pressure breath followed by an increase in cardiac preload during the expiration of a positive pressure breath 9,10. Using this change in arterial pressure, information about cardiac preload or volume status can be inferred. The most common forms of dynamic pressure monitoring that are used are systolic pressure variation and pulse pressure variation.

Several adult studies have shown that systolic pressure variation (SPV) and pulse pressure variation (PPV) more accurately predict fluid response (defined in majority of studies as increase stroke volume index or cardiac index/output >15% after receiving a fluid bolus) in mechanically ventilated critically ill patients compared to static measures, such as CVP (2,10-24). PPV has also been shown to be predictive of fluid responsiveness in many patients with many different pathologies including intraoperative patients, postoperative cardiac bypass patients, patients in septic shock and patients with acute lung injury requiring lower tidal volumes (11,13-15,17-23,25). PPV has also been validated as a helpful and accurate guide for fluid responsiveness in clinical scenarios requiring vasopressors (12,26). Lopes et al demonstrated not only that PPV accurately predicts fluid response, but by using PPV directed fluid resuscitation in the operating room, patients had better postoperative outcomes as defined by decreased ventilator time (1 vs 5 days, P<0.05), and decreased length of hospital stay (7 vs 17 days, P< 0.1) (22).

There are very few studies evaluating pulse pressure variation in the pediatric patient population and results have been mixed. Similar to the adult studies, these studies evaluated dynamic parameters, including SPV and/or PPV, by comparing changes in dynamic parameters to changes seen in stroke volume index calculated by continuous cardiac index monitoring or echocardiogram. Fluid boluses were given and if the SPV or PPV decreased as the stroke volume index increased, then these dynamic parameters were proven to be predictive of fluid responsiveness. Some studies showed that PPV or SPV were not reliable predictors of fluid responsiveness (27-29). In contrast, a study in infants and neonates undergoing congenital heart surgery (ventricular septal defect and atrial septal defect repairs) illustrated that PPV was predictive of fluid response both before and after repair of the cardiac lesion (30). This study was particularly interesting since PPV was able to predict fluid response in two different physiologic states, with and without an intracardiac shunt (30). Two other pediatric studies also demonstrated that dynamic parameters were predictive of fluid response (31,32). There have been no pediatric studies thus far that have investigated if dynamic variable (PPV or SPV) guided fluid resuscitation improves patient outcomes.

Dynamic pressure monitoring, including PPV and SPV, is considered standard of care within the adult anesthesia setting and is currently being used in the adult operating rooms at University of North Carolina Hospitals. Most of the monitors within the hospital are equipped to measure PPV, including the monitors in the PICU. Several PICU attendings and fellows are familiar with PPV and have been using it as an aid in fluid management over the last couple of months. The investigator's hope is that with the use of PPV that physicians will be better able to gauge a patient's intravascular status and judiciously give fluid leading to appropriate fluid management and better patient outcomes in the Pediatric Intensive Care Unit (PICU).

Hypothesis: Using pulse pressure variation will reduce the amount of fluid in the first 48 hours of acute illness (first 48 hours after placement of arterial line and intubation on conventional mechanical ventilation) by 30%. Appropriate fluid management will reduce the amount of time on the ventilator, the number of days in the PICU, and time on vasopressors.

Methods:

Patient Population and Recruitment: All patients admitted to the pediatric intensive care unit will be screened for recruitment for study by pediatric critical care attending or fellow. Patients that require standard mechanical ventilation and arterial line will be eligible for the study. Study will include 75 patients admitted to the PICU that require an arterial line and conventional mechanical ventilation that will be prospectively followed. There will be 75 matched, historic patients that will be used for controls. The investigators do not expect any difficulty enrolling 75 patients to the study as there were 1069 patients admitted to the PICU in the last year (July 2013 to July 2014).

Study Procedure: Prior to any accrual of patients, all nurses in the PICU and all PICU physicians (attendings and fellows) will have formal education and training on use of PPV and the study protocol. In addition, all physicians will have consent training. All patients admitted to the pediatric intensive care unit who are mechanically ventilated on conventional ventilator settings with arterial line will be eligible for the study. Primary investigator (during the day) or physician on call in the PICU (during the night) will obtain consent if patient is eligible for the study. The bedside physician (co-investigator) will give fluid as needed based on standard clinical data (heart rate, central venous pressure if available, blood pressure, urine output, physical exam, lactate level) and pulse pressure variation. Boluses of 5 cc/kg will be given so as to give fluid incrementally. Pulse pressure variation value before fluid bolus and after fluid bolus will be recorded in the electronic medical record. Pulse pressure variation will be followed for 48 hours. Pulse pressure variation, central venous pressure, total fluid for PICU stay, total fluid during 48 hours while on the PPV protocol (cc/kg/day), days mechanically ventilated, hours on vasopressors, any echocardiograms, age, weight at admission, daily weights, sex, diagnosis will be recorded in the patient's medical record. All data will be collected from patient's record by the primary investigator.

Data Analysis: Continuous baseline variables will have descriptions with means and standard deviations, and categorical baseline variables will be described with frequency distributions. A two-sided t-test and corresponding confidence interval will be used to compare matched historic controls to prospectively recruited test group subjects for total amount of fluid in 48 hours (cc/kg/day). Wilcoxon Rank Sum tests for time-to-event data will be applied to time on ventilator (days), time in the PICU (days), and time on vasopressors (hours), together with Kaplan-Meyer curves for descriptive purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to the University of North Carolina pediatric critical care unit, includes all patients admitted to the pediatric critical care service as well as all post-operative patients.
2. No limitations for age or gender.
3. Patient requires standard mechanical ventilation.
4. Patient has an arterial line in place.

Exclusion Criteria:

1. Patient not mechanically ventilated.
2. Patient does not have arterial line placed.
3. Patient requires extracorporeal life support.
4. Patient requires placement on high frequency oscillatory ventilation.
5. Pulse pressure variation unable to be obtained on monitor.
6. Patient has open chest.
7. Patient has arrhythmias.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R Hines, MD, Principal Investigator — University of North Carolina; Umesh Joashi, MD, Study Director — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brierley J, Carcillo JA, Choong K, Cornell T, Decaen A, Deymann A, Doctor A, Davis A, Duff J, Dugas MA, Duncan A, Evans B, Feldman J, Felmet K, Fisher G, Frankel L, Jeffries H, Greenwald B, Gutierrez J, Hall M, Han YY, Hanson J, Hazelzet J, Hernan L, Kiff J, Kissoon N, Kon A, Irazuzta J, Lin J, Lorts A, Mariscalco M, Mehta R, Nadel S, Nguyen T, Nicholson C, Peters M, Okhuysen-Cawley R, Poulton T, Relves M, Rodriguez A, Rozenfeld R, Schnitzler E, Shanley T, Kache S, Skippen P, Torres A, von Dessauer B, Weingarten J, Yeh T, Zaritsky A, Stojadinovic B, Zimmerman J, Zuckerberg A. Clinical practice parameters for hemodynamic support of pediatric and neonatal septic shock: 2007 update from the American College of Critical Care Medicine. Crit Care Med. 2009 Feb;37(2):666-88. doi: 10.1097/CCM.0b013e31819323c6. PMID 19325359
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Boyd JH, Forbes J, Nakada TA, Walley KR, Russell JA. Fluid resuscitation in septic shock: a positive fluid balance and elevated central venous pressure are associated with increased mortality. Crit Care Med. 2011 Feb;39(2):259-65. doi: 10.1097/CCM.0b013e3181feeb15. PMID 20975548
- [Background] Rosenberg AL, Dechert RE, Park PK, Bartlett RH; NIH NHLBI ARDS Network. Review of a large clinical series: association of cumulative fluid balance on outcome in acute lung injury: a retrospective review of the ARDSnet tidal volume study cohort. J Intensive Care Med. 2009 Jan-Feb;24(1):35-46. doi: 10.1177/0885066608329850. Epub 2008 Dec 22. PMID 19103612
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] Marik PE, Cavallazzi R. Does the central venous pressure predict fluid responsiveness? An updated meta-analysis and a plea for some common sense. Crit Care Med. 2013 Jul;41(7):1774-81. doi: 10.1097/CCM.0b013e31828a25fd. PMID 23774337
- [Background] Tibby SM, Hatherill M, Marsh MJ, Murdoch IA. Clinicians' abilities to estimate cardiac index in ventilated children and infants. Arch Dis Child. 1997 Dec;77(6):516-8. doi: 10.1136/adc.77.6.516. PMID 9496187
- [Background] Egan JR, Festa M, Cole AD, Nunn GR, Gillis J, Winlaw DS. Clinical assessment of cardiac performance in infants and children following cardiac surgery. Intensive Care Med. 2005 Apr;31(4):568-73. doi: 10.1007/s00134-005-2569-5. Epub 2005 Feb 15. PMID 15711976
- [Background] Perel A, Pizov R, Cotev S. Respiratory variations in the arterial pressure during mechanical ventilation reflect volume status and fluid responsiveness. Intensive Care Med. 2014 Jun;40(6):798-807. doi: 10.1007/s00134-014-3285-9. Epub 2014 Apr 16. PMID 24737260
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Hadian M, Severyn DA, Pinsky MR. The effects of vasoactive drugs on pulse pressure and stroke volume variation in postoperative ventilated patients. J Crit Care. 2011 Jun;26(3):328.e1-8. doi: 10.1016/j.jcrc.2010.08.018. Epub 2010 Oct 30. PMID 21036528
- [Background] Preisman S, Kogan S, Berkenstadt H, Perel A. Predicting fluid responsiveness in patients undergoing cardiac surgery: functional haemodynamic parameters including the Respiratory Systolic Variation Test and static preload indicators. Br J Anaesth. 2005 Dec;95(6):746-55. doi: 10.1093/bja/aei262. PMID 16286349
- [Background] Huang CC, Fu JY, Hu HC, Kao KC, Chen NH, Hsieh MJ, Tsai YH. Prediction of fluid responsiveness in acute respiratory distress syndrome patients ventilated with low tidal volume and high positive end-expiratory pressure. Crit Care Med. 2008 Oct;36(10):2810-6. doi: 10.1097/CCM.0b013e318186b74e. PMID 18766099
- [Background] Yazigi A, Khoury E, Hlais S, Madi-Jebara S, Haddad F, Hayek G, Jabbour K. Pulse pressure variation predicts fluid responsiveness in elderly patients after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):387-90. doi: 10.1053/j.jvca.2011.09.014. Epub 2011 Nov 17. PMID 22100211
- [Background] Pizov R, Segal E, Kaplan L, Floman Y, Perel A. The use of systolic pressure variation in hemodynamic monitoring during deliberate hypotension in spine surgery. J Clin Anesth. 1990 Mar-Apr;2(2):96-100. doi: 10.1016/0952-8180(90)90061-7. PMID 2346658
- [Background] Cannesson M, Slieker J, Desebbe O, Bauer C, Chiari P, Henaine R, Lehot JJ. The ability of a novel algorithm for automatic estimation of the respiratory variations in arterial pulse pressure to monitor fluid responsiveness in the operating room. Anesth Analg. 2008 Apr;106(4):1195-200, table of contents. doi: 10.1213/01.ane.0000297291.01615.5c. PMID 18349192
- [Background] Auler JO Jr, Galas F, Hajjar L, Santos L, Carvalho T, Michard F. Online monitoring of pulse pressure variation to guide fluid therapy after cardiac surgery. Anesth Analg. 2008 Apr;106(4):1201-6, table of contents. doi: 10.1213/01.ane.0000287664.03547.c6. PMID 18349193
- [Background] Derichard A, Robin E, Tavernier B, Costecalde M, Fleyfel M, Onimus J, Lebuffe G, Chambon JP, Vallet B. Automated pulse pressure and stroke volume variations from radial artery: evaluation during major abdominal surgery. Br J Anaesth. 2009 Nov;103(5):678-84. doi: 10.1093/bja/aep267. Epub 2009 Sep 29. PMID 19797246
- [Background] Kramer A, Zygun D, Hawes H, Easton P, Ferland A. Pulse pressure variation predicts fluid responsiveness following coronary artery bypass surgery. Chest. 2004 Nov;126(5):1563-8. doi: 10.1378/chest.126.5.1563. PMID 15539728
- [Background] Michard F, Boussat S, Chemla D, Anguel N, Mercat A, Lecarpentier Y, Richard C, Pinsky MR, Teboul JL. Relation between respiratory changes in arterial pulse pressure and fluid responsiveness in septic patients with acute circulatory failure. Am J Respir Crit Care Med. 2000 Jul;162(1):134-8. doi: 10.1164/ajrccm.162.1.9903035. PMID 10903232
- [Background] Lopes MR, Oliveira MA, Pereira VO, Lemos IP, Auler JO Jr, Michard F. Goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery: a pilot randomized controlled trial. Crit Care. 2007;11(5):R100. doi: 10.1186/cc6117. PMID 17822565
- [Background] Freitas FG, Bafi AT, Nascente AP, Assuncao M, Mazza B, Azevedo LC, Machado FR. Predictive value of pulse pressure variation for fluid responsiveness in septic patients using lung-protective ventilation strategies. Br J Anaesth. 2013 Mar;110(3):402-8. doi: 10.1093/bja/aes398. Epub 2012 Nov 15. PMID 23161359
- [Background] Michard F, Chemla D, Richard C, Wysocki M, Pinsky MR, Lecarpentier Y, Teboul JL. Clinical use of respiratory changes in arterial pulse pressure to monitor the hemodynamic effects of PEEP. Am J Respir Crit Care Med. 1999 Mar;159(3):935-9. doi: 10.1164/ajrccm.159.3.9805077. PMID 10051276
- [Background] Pizov R, Ya'ari Y, Perel A. Systolic pressure variation is greater during hemorrhage than during sodium nitroprusside-induced hypotension in ventilated dogs. Anesth Analg. 1988 Feb;67(2):170-4. PMID 3341566
- [Background] Byon HJ, Lim CW, Lee JH, Park YH, Kim HS, Kim CS, Kim JT. Prediction of fluid responsiveness in mechanically ventilated children undergoing neurosurgery. Br J Anaesth. 2013 Apr;110(4):586-91. doi: 10.1093/bja/aes467. Epub 2012 Dec 18. PMID 23250892
- [Background] Saxena R, Durward A, Puppala NK, et al. A comparison between novel static and dynamic markers of fluid responsiveness: preliminary data from 47 children. Proc 22nd Annu Congr ESPNIC. 2011;37 Suppl 2:S315-442. doi:10.1007/s00134-011-2387-x.
- [Background] Pereira de Souza Neto E, Grousson S, Duflo F, Ducreux C, Joly H, Convert J, Mottolese C, Dailler F, Cannesson M. Predicting fluid responsiveness in mechanically ventilated children under general anaesthesia using dynamic parameters and transthoracic echocardiography. Br J Anaesth. 2011 Jun;106(6):856-64. doi: 10.1093/bja/aer090. Epub 2011 Apr 26. PMID 21525016
- [Background] Renner J, Broch O, Duetschke P, Scheewe J, Hocker J, Moseby M, Jung O, Bein B. Prediction of fluid responsiveness in infants and neonates undergoing congenital heart surgery. Br J Anaesth. 2012 Jan;108(1):108-15. doi: 10.1093/bja/aer371. Epub 2011 Nov 23. PMID 22113930
- [Background] McLean JRL, Inwald DP. The utility of stroke volume variability as a predictor of fluid responsiveness in critically ill children: a pilot study. Intensive Care Med. 2014 Feb;40(2):288-289. doi: 10.1007/s00134-013-3171-x. Epub 2013 Dec 5. No abstract available. PMID 24306083
- [Background] Lee JY, Kim JY, Choi CH, Kim HS, Lee KC, Kwak HJ. The ability of stroke volume variation measured by a noninvasive cardiac output monitor to predict fluid responsiveness in mechanically ventilated children. Pediatr Cardiol. 2014 Feb;35(2):289-94. doi: 10.1007/s00246-013-0772-7. Epub 2013 Aug 21. PMID 23963186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective subjects were considered for enrollment if less than 17 years of age and admitted to the pediatric critical care unit. In addition subjects had to require conventional mechanical ventilation and have an arterial line. Prospective recruitment time between 11/26/2014 and 3/1/2016.
Pre-assignment Details: Prospective subjects per the protocol were allowed more than one enrollment on the study during the same admission once recruited. There were 46 unique prospective subjects with 50 enrollments and 50 retrospective enrollments. Numbers below and throughout the results section represent number of enrollments or participation.
Groups:
- Prospective: Patients in this arm will have fluid given based on standard clinical data (blood pressure, heart rate, lactate level, urine output, clinical exam) in addition to information provided by automated pulse pressure variation (PPV). PPV will be followed for first 48 hours after recruitment to the study. Fluid (normal saline, albumin 5%, hetastarch per the clinician preference) will be given in 5ml/kg increments for PPV> 13.
  Automated Pulse Pressure Variation: Based on standard of care, the physician will give fluid as needed based on standard clinical data (heart rate, central venous pressure if available, blood pressure, urine output, physical exam, lactate level) and pulse pressure variation. PPV should be elevated consistently greater than 15 minutes before giving fluid without other symptoms of patient instability (low blood pressure, elevated lactate, tachycardia). Pulse pressure variation will be followed for 48 hours.
- Retrospective: Patients in this arm were previously admitted to the PICU and were given fluid based on standard clinical data (blood pressure, heart rate, lactate level, urine output, clinical exam). PPV was not used to guide therapy in this group of patients.
Period: Overall Study
Arm/Group | Prospective | Retrospective
Started | 50 (Started enrollment and recruitment 11/26/2014) | 50 (Consider eligible for retrospective enrollment if admitted after 4/1/2012)
Completed | 50 (Ended enrollment and recruitment 3/1/2016) | 50 (Consider eligible for retrospective enrollment if admitted up until 10/15/2012)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects admitted to the pediatric critical care unit
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective | Retrospective | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.099 (5.765) | 4.144 (5.828) | 4.121 (5.738)
Gender [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 31 | 23 | 54
Diagnosis [Number; unit: participants]
  Primary Respiratory Failure | 7 | 7 | 14
  Sepsis | 7 | 7 | 14
  Diabetic Ketoacidosis | 1 | 1 | 2
  Persistent Pulmonary Hypertension of the Newborn | 1 | 1 | 2
  Neuroblastoma | 1 | 1 | 2
  Spinal Fusion | 4 | 4 | 8
  Craniotomy | 1 | 1 | 2
  Congenital Diaphragmatic Hernia | 2 | 2 | 4
  Congenital Cardiac Disease | 24 | 24 | 48
  Cerebral Edema | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Fluid (ml/kg/Day) Given
Description: Total fluid (ml/kg/day) given during the first 48 hours of enrollment
Time Frame: First 48 hours after enrollment
Measure: Mean (Standard Deviation); unit: ml/kg/day
Groups:
- Prospective: Patients in this arm will have fluid given based on standard clinical data (blood pressure, heart rate, lactate level, urine output, clinical exam) in addition to information provided by automated pulse pressure variation (PPV).
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 50 | 50
ml/kg/day | 124.38 (63.05) | 122.099 (50.27)

2. Primary Outcome: Total Fluid Bolused
Description: Total fluid bolused within 48 hours after enrollment.
Time Frame: 48 hours after enrollment
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 50 | 50
ml/kg | 11.55 (16.34) | 28.08 (56.60)

3. Secondary Outcome: Number of Hours on Vasopressors
Description: Hours that a subject remained intubated during pediatric intensive care admission during subject recruitment
Time Frame: From pediatric ICU admission to pediatric ICU discharge (up to 149 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 50 | 50
hours | 71.74 (123) | 42.4 (63.2)

4. Secondary Outcome: Number of Days on Ventilatory Support
Description: Number of days subject was on ventilatory support (during time of subject enrollment) to the pediatric critical care unit. This included subjects that were intubated or was on a ventilator with a tracheotomy
Time Frame: From pediatric ICU admission to pediatric ICU discharge (up to 149 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 50 | 50
days | 23.8 (45.6) | 8.68 (9.7)

5. Secondary Outcome: Number of Days in the PICU
Description: Number of days for admission pediatric critical care unit (admission during which subject was enrolled into the study)
Time Frame: From pediatric ICU admission to pediatric ICU discharge (up to 149 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 50 | 50
days | 28.66 (36.64) | 12.48 (11.85)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded until subjects discharge from the pediatric critical care unit.
Description: There was no recording or evaluation of adverse events in the retrospective group since they were evaluated retrospectively. The adverse events recorded are more likely secondary to the critically ill nature of the cohort rather than PPV itself.
Arm/Group | Prospective | Retrospective
Serious Adverse Events (participants affected / at risk) | 22/50 | 0/0
Other Adverse Events (participants affected / at risk) | 0/50 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective (N=50) | Retrospective (N=0)
Death (Investigations) | 5 (5) | 0 (0) — Patients that died during the time enrolled in the study or until discharge from the pediatric critical care unit.
Extracorporeal Life Support (Investigations) | 2 (2) | 0 (0) — Subjects requiring extracorporeal life support during time of study or during enrolled admission to the pediatric critical care unit.
Prolonged Intubation (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 0 (0) — Subject requiring intubation longer that expected course during enrolled admission in the pediatric critical care unit
Fluid Overload (Renal and urinary disorders) | 3 (3) | 0 (0) — Subjects that had significant fluid overload requiring significant, unexpected diuresis or hemodialysis
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0) — Subject with renal failure significant enough to require hemodialysis or peritoneal dialysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No